CLINICAL TRIAL: NCT03435653
Title: Comparative Clinical and Radiographic Evaluation of Demineralized Freeze-dried Bone Allograft With and Without Decortication in the Treatment of Periodontal Intrabony Defects - a Randomized Controlled Clinical Study.
Brief Title: Regenerative Therapy of Periodontal Bone Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amanpreet Periodontics
Record Dates: First submitted 2018-02-01; First posted 2018-02-19 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-01

CONDITIONS: Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Cerebral Decortication; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group OFD with DFDBA
  Interventions: Other: OFD with DFDBA
- Test group (Experimental): Test group OFD with decortication and DFDBA
  Interventions: Other: OFD with decortication and DFDBA

INTERVENTIONS:
Other: OFD with DFDBA — Control Group Open flap debridement with DFDBA Periodontal surgery will be performed in the form of open flap debridement along with placement of demineralized freeze dried bone allograft at the defect site.
  Other Names: regenerative material and periodontal surgery
  Arms: Control group
Other: OFD with decortication and DFDBA — Test Group Open flap debridement with decortication and demineralised freeze dried bone allograft Open flap debridement with decortication and placement of demineralized freeze dried bone allograft at the defect site.
  Other Names: regenerative material ,decortication with surgery
  Arms: Test group

SUMMARY:
To compare clinically and radiographically the efficacy of demineralized freeze-dried bone allograft with and without decortication in the treatment of periodontal intrabony defects assessed by gain in clinical attachment, reduction of pocket depth and radiographic bone fill.To evaluate clinically and radiographically the regenerative potential of demineralized freeze-dried bone graft (DFDBA) material in periodontal intrabony defects.To evaluate clinically and radiographically the regenerative potential of demineralized freeze-dried bone graft (DFDBA) when used in combination with decortication in periodontal intrabony defects.

DETAILED DESCRIPTION:
INTRODUCTION Periodontitis is a multifactorial infectious disease with microbial plaque as initiator that triggers inflammatory response in the periodontal tissue. As the disease progresses, symptoms may include bleeding gums, periodontal abscesses, increased tooth mobility due to the loss of bone support, tooth migration, exposure of the root surface, and tooth loss. Current periodontal therapy is directed towards establishing a healthy periodontium by attempting to resolve the tissue inflammation induced by bacterial plaque and its products and the restitution of the anatomic defects caused by the disease process. There are many outcomes possible from the periodontal therapy depending upon the goals, the type of therapy, and the methods utilized to evaluate it. These can range from halting the destructive process, maintaining an area to repair a defect and/or regeneration.

Melcher described the concept of selective cell repopulation of defects to enhance healing.The guided tissue regeneration (GTR) technique excludes faster growing epithelial and connective tissue cells with barriers and bone grafts to allow slower moving pluripotential and osteogenic cells to repopulate the treated site. To attain horizontal and/or vertical bone augmentation beyond the envelope of skeletal bone, four principles need to be met: primary wound closure, angiogenesis to provide necessary blood supply and undifferentiated mesenchymal cells, space maintenance and stability of the blood clot .The ultimate goal of the regenerative periodontal therapy is to restore the lost periodontal tissues including cementum, periodontal ligament and alveolar bone.

The current regenerative therapy includes the use of bone grafts, guided tissue regeneration (GTR), bioactive agents like Enamel matrix derivative (EMD) and laser assisted regeneration. The clinical periodontal regenerative treatments focus on the utilization of bone grafts that can be obtained from the same individual (autografts), from different individual of the same species (allografts) or from a different species (xenografts). Apart from these synthetic bone grafts are also available (alloplasts).

Allografts are bone grafts taken for transplantation from one human to another. There are two types of allografts available including freeze-dried bone allograft and demineralized freeze-dried bone allograft (DFDBA). Demineralized freeze-dried bone allograft is a graft that possesses osteoconductive and osteoinductive properties. Demineralization process of the graft exposes the bone inductive properties located in the bone matrix such as bone morpogenetic protein-2(BMP2) and bone morpogenetic protein-7 (BMP 7) that aid in mesenchymal cell migration, attachment and osteogenesis when implanted in well vascularised bone. It has shown to regenerate bone as well as cementum and periodontal ligament in treatment of periodontal osseous defects at the same time eliminates the need for a second surgical site. When used for periodontal regeneration, DFDBA may not only lead to clinical improvements in terms of pocket probing depth (PPD) reduction and gain of clinical attachment level (CAL), but also lead to formation of new connective tissue attachment and new alveolar bone.

Several authors have advocated the use intramarrow penetration (IMP), also known as decortication, as a part of guided bone regeneration procedure. Osteoblasts that form new bone are derived from periosteum, endosteum, and undifferentiated pluripotential mesenchymal cells in the bone marrow. After the elevation of mucoperiosteal flap when the barrier is placed, the contribution of periosteum to GBR procedure is lost. Along with this, a bone graft placed on the cortical bone also interferes with the entry of undifferentiated pluripotential mesenchymal cells from the endosteum and bone marrow towards the GBR-treated site.Therefore drilling holes through cortical bone into more vascular cancellous bone induces bleeding and organised clot releases cytokines and growth factors which attracts the blood vessels, osteoblasts, and pluripotential cells to the grafted sites. It also enhance the physical connection between the bone graft and recipient site to improve its stability and provide firm linking for newly generated bone.Studies have shown that open flap debridement (OFD) combined with decortication produces positive result outcomes in regenerative periodontal treatment.

It is hypothesized that placement of demineralized freeze dried bone allograft along with decortication would provide predictable periodontal regeneration as compared to placement of demineralized freeze dried bone allograft alone in 2-,3- or combined 2,3 wall intrabony defects. Therefore to support or reject the hypothesis, this study will be conducted to evaluate the periodontal parameters in terms of periodontal healing by regenerative periodontal therapy with demineralized freeze dried bone allograft with and without decortication in the treatment of 2-, 3- or combined 2,3 wall periodontal defects .

MATERIALS AND METHOD STUDY POPULATION AND DESIGN The study will be conducted in the department of Periodontics and Oral Implantology at Pandit B.D.Sharma university of health sciences, Rohtak according to the 1975 Helsinki Declaration, as revised in 2013.

This interventional study will include systemically healthy minimum 36 patients with 2-, 3-or 2,3 wall periodontal intrabony defects which will be equally divided into two groups. Individuals will be selected randomly, with no discrimination on the basis of caste, sex, religion or socio-economic status.

Per patient one defect will be selected and deepest intrabony defect will be considered.

Control Group Open flap debridement with DFDBA:Periodontal surgery will be performed in the form of open flap debridement along with placement of demineralized freeze dried bone allograft at the defect site.

Test Group Open flap debridement with decortication and demineralised freeze dried bone allograft:Open flap debridement with decortications and placement of demineralized freeze dried bone allograft at the defect site.

CLINICAL PARAMETERS Full mouth indices to be recorded at baseline Bleeding on probing Probing Pocket depth Clinical Attachment loss Site specific indices Plaque index (PI) Silness and Loe 1964. Gingival index (GI) Loe H and Silness 1963. Probing Pocket depth (PPD)will be measured as mm distance from gingival margin to the base of pocket.

Clinical attachment loss (CAL) will be measured as distance from cemento-enamel junction to the base of pocket.

Bleeding on probing (BOP) Tooth mobility Gingival recession (REC) measurement will be made by periodontal probe from cemento-enamel junction to the gingival crest.

Keratinized tissue width (KTW) distance from the gingival margin to the mucogingival junction.

Using UNC 15 periodontal probe to measure PPD, CAL, BOP, gingival recession at 6 sites (mesial, distal, median points at buccal and lingual aspects) per tooth and at 4 sites per tooth to measure PI, GI.The cemento-enamel junction will be used as a fixed reference point.

RADIOGRAPHIC PARAMETERS Customized bite blocks and parallel angle technique will be used to obtain Intraoral Periapical radiographs. Following parameters should be assessed and will be measured using imaging software.

Radiographic defect depth (rDD) defined as the distance from the projection on the root surface of the most coronal point of the residual bone crest to the bottom of the defect.

Radiographic defect width (rDW)defined as the distance from the most coronal point of the residual bone crest to the root surface, were measured using a caliper and recorded to the nearest mm.

Radiographic defect angle (ANG)defined by a line tangential to the root surface and a line connecting the bottom of the defect to the most coronal part of the crest next to the adjacent tooth.

Recall appointments will be scheduled weekly during the first postoperative month;3 month, 6 month and 9 month interval. All clinical parameters and radiographic parameters will be recorded at baseline, 6 month and 9 month post surgery. The cemento-enamel junction(CEJ) will be used as a fixed reference point.

METHODOlLOGY PRESURGICAL THERAPY includes Oral hygiene instructions Full mouth supragingival and subgingival scaling and root planning with ultrasonic scaler, hand scaler and curettes.

Patient will be recalled after 6 weeks, during which his/her oral hygiene status will be checked. Patients with low levels of residual infection (Full-Mouth Bleeding Score FMBS < 20%) and good oral hygiene status (Plaque Index- <1[Silness and loe]) will be considered for further surgery.

PERIODONTAL SURGICAL PROCEDURE After administration of local anaesthesia, buccal and lingual/palatal intracrevicular incision will be made and mucoperiosteal flaps will be reflected including atleast one tooth ahead and another behind the treated tooth. Meticulous defect debridement and root planning will be carried out using area specific curettes and scalers. After instrumentation, the root surfaces will be irrigated with saline solution in attempt to remove any remaining detached fragments from the defect and surgical field.

The following clinical parameters will be then recorded at the deepest point: CEJ to alveolar bone crest (CEJ-BC); CEJ to surgical bottom of the defect (CEJ-sBD); defect depth (BC-sBD); defect width (DW), distance from root surface to most coronal extension of alveolar crest and number of defect walls.

In the control group, DFDBA is placed at the defect site and mucoperiosteal flaps will be repositioned and secured by 3-0 non absorbable black silk surgical suture whereas in the test group, the intrabony defect cortical walls will be penetrated using a round carbide bur (1mm diameter) to reach the marrow space and then demineralized freeze dried bone allograft is placed at the defect site. Flap will be closed in the same manner as in the control group.

The surgical area will be protected and covered with periodontal dressing and post operative instructions will be given.

ELIGIBILITY:
Inclusion Criteria:

* Age-28-60 years , patients with chronic periodontitis according to criteria of Armitage GC classification system for periodontal diseases and conditions32.
* Presence of 2-, 3-, or combined 2-3-wall intrabony defect ≥ 3 mm deep assessed by transgingival probing and intraoral periapical radiograph, to be confirmed after flap elevation.
* Test tooth and adjoining teeth testing vital, should be free of caries or inadequate restorations.
* Non smokers
* Completed etiological periodontal therapy (oral hygiene instructions and scaling and root-planing with Full-Mouth Bleeding Score FMBS < 20% and plaque index score<1 [Silness and Loe 1964]33).

TOOTH OR DEFECT ELIGIBILITY CRITERIA-

* 2-, 3- or combined 2,3-wall intrabony defect.
* Pocket probing depth ≥ 5 mm
* CAL ≥ 5 mm.
* Tooth mobility < grade 1

Exclusion Criteria:

* Systemic illness known to affect the periodontium or outcome of periodontal therapy.
* Patient taking medications such as corticosteroids or calcium channel blockers, which are known to interfere periodontal wound healing or patient on long term NSAID therapy.
* Patient allergic to study medications
* Pregnant or lactating mothers.
* Tooth with 1wall intrabony defect.
* Grade2, grade 3 mobile teeth.
* Defects extending to a root furcation area.
* Unrestorable tooth.
* Fractured/perforated roots.
* Developing permanent tooth.
* Endodontically treated tooth.
* Presence of non working interferences.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Radiographic Bone fill | 12 months
  gain in bone level in mm
CAL | 12 months
  clinical attachment level in mm

CONTACTS AND LOCATIONS:
Overall Officials: Amanpreet Kaur, Principal Investigator — Post Graduate Institute of Dental Sciences, Rohtak
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India